CLINICAL TRIAL: NCT03902405
Title: CEASAR (Computerized Exercise to Alter Stimulant Approach Responses) - Piloting a Novel Intervention to Improve Outcomes in Individuals Suffering From Cocaine or Methamphetamine Use Disorder: A Randomized Controlled Study
Brief Title: Computerized Exercise to Alter Stimulant Approach Responses
Acronym: CEASAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christian Schutz, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H16-01099
Record Dates: First submitted 2019-03-27; First posted 2019-04-04 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Amphetamine-Related Disorders; Cocaine-Related Disorders; Substance-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders; Cocaine-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active CEASAR Intervention (Active Comparator): Participants will be given the active CEASAR intervention where they will be trained to "avoid" cues associated with stimulant use and approach healthy cues based on the orientation of the images presented. Individuals will be asked to approach (pull in) portrait images and avoid (push away) landscape images. In the active condition, pushed pictures (landscape orientation) will exclusively be stimulant-use related pictures. Conversely, healthy images will be in the portrait orientation which will be pulled in.
  Interventions: Behavioral: Active CEASAR Intervention
- Placebo CEASAR (Placebo Comparator): In the control condition, stimulant use-related pictures will be randomized and equally divided into push (landscape) and pull (portrait) conditions.
  Interventions: Behavioral: Placebo CEASAR

INTERVENTIONS:
Behavioral: Active CEASAR Intervention — Healthy and stimulant-use related pictures will be presented on a computer screen. Using a joystick, participants will be trained to pull in pictures that are presented in portrait orientation, and push those presented horizontally. In the active experimental condition, pushed pictures will exclusively be stimulant-related pictures.
  Arms: Active CEASAR Intervention
Behavioral: Placebo CEASAR — In the control condition, stimulant cues and healthy cues will be randomized and stimulant use-related pictures will be equally divided into push and pull conditions.
  Arms: Placebo CEASAR

SUMMARY:
The purpose of this study is to evaluate the Computerized Exercise to Alter Stimulant Approach Responses (CEASAR), a novel stimulant use cessation intervention, for clients currently enrolled in a treatment centre for mental health and addiction. The investigators plan to conduct a randomized, single-blind controlled trial involving inpatients presenting with concurrent disorders to test the impact of this novel computerized intervention. This pilot study will be conducted at the Burnaby Centre for Mental Health and Addiction (BCMHA) in Burnaby, BC, Canada.

DETAILED DESCRIPTION:
Purpose: To examine a novel computerized exercise intervention as an add-on to currently available evidence-based stimulant use cessation treatments. This study will evaluate whether or not this intervention can improve stimulant use disorder outcomes in a population with concurrent disorders that are difficult to treat.

Hypothesis: 1) The intervention will be easy to integrate in the existing program. 2) Participation in the experimental (stimulant-avoidance) condition will reduce craving (as assessed by the stimulant craving questionnaire brief version), show reduction in an automatic association of activities with stimulant use and stimulant relapses (as assessed by behaviour association questionnaires) and have reduced relapses as assessed by urine drug screens in 12 weeks following initiation of the intervention.

Justification: Stimulant use disorders are among the most challenging disorders, specifically in individuals suffering from concurrent disorders or also identified as dual diagnosis. While medication is available to support the treatment of other substance use disorders (alcohol, opioids, tobacco), currently there is none to treat stimulant use disorders, such as cocaine use disorder and methamphetamine use disorder. Recently, a group in Europe developed the "retraining of automatic approach" intervention, which is based on simple mechanistic retraining for avoidance of substances. This method was successfully applied to change drinking behaviour in a sample of alcoholic inpatients. Participants respond to substance cues by initiating a distancing activity (pushing a joystick away). In contrast, healthy activities are "approached" or pulled in using the joystick. This differential activity trains participants to alter initial responses and "cognitive biases" to simply and automatically avoid substances.

Objectives: Test the hypothesis and evaluate whether or not the Computerized Exercise to Alter Stimulant Approach Responses (CEASAR) can improve stimulant use disorder outcomes in a population with concurrent disorders that are difficult to treat.

Research design: This study is a randomized, single blind, controlled trial involving in-patients with a stimulant use disorder. The participants will be split up equally into 2 groups: the active CEASAR intervention (experimental condition) and the placebo intervention (control). Patients are able to stay at the BCMHA for 6 months with the average being 4-5 months and the study will take place over 12 weeks during their stay. Both groups will use a joystick to push away ("avoid") or pull in ("approach") randomized stimulant and healthy cues presented on a computer screen. In the experimental condition, pushed pictures will exclusively be stimulant use-related pictures, while pulled pictures will be exclusively healthy. In the control condition, stimulant use-related pictures will be equally divided into push and pull conditions. Some of the cues will be visual (e.g. pictures of cocaine powder, pipes, needles etc.) and some of them will be textual (e.g. words like eight ball, rock, etc.).

ELIGIBILITY:
Inclusion Criteria:

* In-patient of the Burnaby Centre of Mental Health & Addiction
* 19 years of age or older
* Individuals with a current stimulant use disorder (cocaine, crack cocaine, amphetamine, methamphetamine, crystal meth), active before intake at BCMHA (as assessed by the MINI)
* Proficiency to read and write English and competent to provide consent

Exclusion Criteria:

* Individuals not stabilized enough to allow for regular participation in the intervention (determined by treating psychiatrist)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in craving as assessed by the Stimulant Craving Questionnaire-Brief (SCQ-B) | Baseline, 4 weeks, 8 weeks, 12 weeks
  Changes in craving will be assessed at baseline before the intervention, and at 4, 8, and 12 weeks after. It will be assessed by the Stimulant Craving Questionnaire-Brief (SCQ-B), which uses a 7-item scale (0 = Strongly Disagree, 6 = Strongly Agree) that can produce a composite score between 0 and 6. On this scale, lower scores indicate less craving which is considered a better outcome. Higher scores indicate more craving which is considered a worse outcome.
Change in Behavioural association as assessed by the Behaviour Association Scale | Baseline, 4 weeks, 8 weeks, 12 weeks
  The Behaviour Association Scale measures association of substance use with different situations.
  Subscale 1, Word Associations: participants list the first word or phrase they associate with a given word. There are 13 word prompts, so the scale runs from 0 (no prompts associated with substance use) to 13 (all prompts associated with substance use). A low score is considered a better outcome because it means fewer situations are associated with substance use.
  Subscale 2, Behavioral Associations: operates the same way, except that there are 20 prompts listed so the scale runs from 0-20.
  These subscales are each measured on 2 dimensions, for a total of 4 dimensions to the scale.
  Dimension A: Each subscale is self-coded by the participant, where the participant determines if their response is substance-use related. Dimension B: Each subscale is researcher-coded, where 2 coders determine whether or not the response is unambiguously related to substance use.
Relapse to use as assessed by weekly self-reports and urine drug screens | Between week 2 and week 12
  Number of relapse days between week 2 and week 12 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schutz, MD PhD MPH, Principal Investigator — University of British Columbia
Locations (1):
- Burnaby Centre for Mental Health and Addiction, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiers RW, Eberl C, Rinck M, Becker ES, Lindenmeyer J. Retraining automatic action tendencies changes alcoholic patients' approach bias for alcohol and improves treatment outcome. Psychol Sci. 2011 Apr;22(4):490-7. doi: 10.1177/0956797611400615. Epub 2011 Mar 9. PMID 21389338
- [Background] Wiers RW, Rinck M, Kordts R, Houben K, Strack F. Retraining automatic action-tendencies to approach alcohol in hazardous drinkers. Addiction. 2010 Feb;105(2):279-87. doi: 10.1111/j.1360-0443.2009.02775.x. PMID 20078486

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT03902405/Prot_SAP_000.pdf